CLINICAL TRIAL: NCT07034443
Title: Functional Outcomes in Ulcerative Colitis Patients With Ileal Pouch Anal Anastomosis Treated With High Intensity Focused Electromagnetic Stimulation: A Prospective Pilot Study
Brief Title: Functional Outcomes in Ulcerative Colitis Patients With Ileal Pouch Anal Anastomosis Treated With High Intensity Focused Electromagnetic Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Karen Zaghiyan, Colon and Rectal Surgeon, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003888
Record Dates: First submitted 2025-05-16; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Fecal Incontinence
Keywords: Ulcerative colitis; Fecal Incontinence; Functional Outcomes; High Intensity Focused Electromagnetic Stimulation; J pouch
MeSH Terms: conditions — Fecal Incontinence; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- High Intensity Focused Electromagnetic Stimulation (Experimental): This will include all the patients within the study who will be receiving the High Intensity Focused Electromagnetic Stimulation
  Interventions: Device: High Intensity Focused Electromagnetic Stimulation

INTERVENTIONS:
Device: High Intensity Focused Electromagnetic Stimulation — Patients will sit on the device, the high intensity for 28 minutes, twice a week for three weeks

SUMMARY:
The purpose of this research is to evaluate functional outcomes in patients with Ulcerative Colitis and IBDU who have received an ileal pouch anal anastomosis (IPAA), commonly referred to as a J pouch, after treatment with the Emsella chair. We will specifically look at fecal incontinence and patient health related quality of life outcomes before, during and after course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years old or older are included.
* Patients who have a J pouch reconstruction due to Ulcerative Colitis or IBDU
* Must be at least 1 year out from J pouch surgery
* Have fecal incontinence

Exclusion Criteria:

* Any records flagged "break the glass" or "research opt out."
* Pediatric Patients <18 years of age
* Did not receive a J pouch
* Patients who received a J pouch for any other indication, including but not limited to Crohn's disease, familial adenosis polyposis
* Have active pouchitis
* Have an active fistula
* If reclassified to de novo Crohn's after surgery
* Have implanted metal devices or medical devices
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Determine if patients have change in overall quality of live, as determined by statistically significant change in Patient Reported Outcomes Measurement Information System 10 Score from baseline | baseline, 1 month and 3 months
  Patient Reported Outcomes Measurement Information System Score (PROMIS 10), scaled from 0-20 evaluate patient overall quality of life. Higher score indicates better health

SECONDARY OUTCOMES:
Determine change in sexual function and satisfaction in patients at treatment determined by Patient Reported Outcomes Measurement Information System Score sexual function scale | baseline, 1 month, 3 months
  Patient Reported Outcomes Measurement Information System Score (PROMIS) sexual function, scored 0-20 to evaluate patient sexual health. Higher score indicates better sexual function
Determine change in fecal incontinence, as determined by change in Wexner scale from baseline | baseline, 1 and 3 months
  The Wexner Scale ranges from 0-20, with 0 being perfect continence and 20 being complete incontinence
Determine if change in pelvic organ dysfunction as determined by IPSS, CRAD- 9, UD16, POPDI | baseline, 1 and 3 months
  POPDI6 (Pelvic Organ Prolapse Distress Inventory). Score 0-20 with higher score reflecting more severe symptoms of pelvic organ dysfunction.
Determine if change in pelvic organ dysfunction as determined by IPSS | baseline, 1 month and 3 months
  IPSS (International Prostate Symptom Score). Scored 0-20. Higher score indicates more severe symptoms of prostate dysfunction
Determine if change in pelvic organ dysfunction as determined by CRAD- 9 | baseline, 1 month and 3 months
  CRAD-8 (Colorectal Anal Distress Inventory 8 ). Higher scores indicate more severity in pelvic organ dysfunction.
Determine if change in pelvic organ dysfunction as determined by UD16 | Baseline, 1 month and 3 months
  UDI6 (Urinary Distress Inventory 6). Score 0-20, higher number indicated more severe symptoms of dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zaghiyan, MD, Principal Investigator — Cedar Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
PI preference

DOCUMENTS (2):
  • Study Protocol (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT07034443/Prot_000.pdf
  • Informed Consent Form (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT07034443/ICF_001.pdf